CLINICAL TRIAL: NCT02407132
Title: Family Model of Diabetes Self-Management Education in the Marshallese Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 203482
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard DSME (Active Comparator): Participants assigned to this arm received standard diabetes self-management education classes offered at community locations, taught by Certified Diabetes Educators (CDEs) in a group/classroom setting.
  Interventions: Behavioral: Standard DSME
- Adapted DSME (Experimental): Participants assigned to this arm received an intervention that includes culturally-adapted DSME with their participating family members in a family/home setting.
  Interventions: Behavioral: Adapted DSME

INTERVENTIONS:
Behavioral: Adapted DSME — Participants assigned to this arm received an intervention that includes culturally-adapted DSME with their participating family members in a family/home setting.
  Arms: Adapted DSME
Behavioral: Standard DSME — Active Comparator: Standard DSME Participants assigned to this arm received standard diabetes self-management education classes offered at community locations, taught by Certified Diabetes Educators (CDEs) in a group/classroom setting.
  Arms: Standard DSME

SUMMARY:
The investigators will conduct a comparative effectiveness evaluation using a randomized control trial design of a culturally adapted family model of Diabetes Self-Management Education (Adapted DSME) compared with Standard DSME within the Marshallese population. The family model will cover the same concepts as the standard format. However, the family model will incorporate culturally-adapted education and recommendations aimed at engaging family members in the management of the primary participant's diabetes, and family members will be invited to fully participate in the study. By contrast, the standard model provides diabetes self- management education to the diabetic participant only, and the participant's family members do not participate in the classes or any other part of the study. Biometric and survey data will be collected pre-intervention, post-intervention, 6 months post-intervention, and 12 months post-intervention. A qualitative debriefing session will be held for each family between the final DSME session and the 6 month post-intervention to obtain qualitative data regarding the participant's perceptions of the intervention and implementation process.

DETAILED DESCRIPTION:
Background and Rationale

The Marshallese population suffers from a significant and disproportionate burden of type 2 diabetes. The rate of type 2 diabetes among the Marshallese is one of the highest of any population group in the world-at least 400% higher than the general US population.1-7 Our systematic review of local, national, and international data found estimates of diabetes in the Marshallese (populations living both in the US and Marshall Islands) ranging from 30% to 50% compared to 8.3% for the US population and 4% worldwide.4-7 Causes for this disparity have not been completely unraveled and are partially embedded in the history of the Marshall Islands. Between 1946 and 1958, the US military tested nuclear weapons on several of the Marshall Islands. People who inhabited the bombed islands and atolls were relocated, but Marshallese living on nearby atolls that were not evacuated experienced nuclear fallout during and after nuclear tests. Because of the nuclear testing, the Atomic Energy Commission lists the Marshall Islands as one of the most contaminated places in the world, and several studies demonstrate ongoing health effects from the nuclear testing.8 The nuclear contamination resulted in significant and long-term changes in diet and lifestyle of the Marshallese.9-12 These changes in diet and lifestyle have contributed to an increased rate of type 2 diabetes.2-5,16-19 The Compact of Free Association between the Republic of the Marshall Islands (RMI) and the US, signed in 1986, permits the US to conduct military activities in the Marshall Islands and also allows Marshallese individuals to come to the US without a visa. The Marshallese population living in the US tripled between 2000 and 2010, with Arkansas having the largest population of Marshallese living outside of the RMI.

Diabetes self-management education (DSME) is an evidence-based model that has been shown to improve glycemic control, reduce diabetic complications, and reduce the cost of managing diabetes. Standard implementation approaches of DSME have not been effective in Marshallese populations, indicating that a unique approach tailored to this population is needed.2-3 Because of the disproportionate burden of diabetes and related complications experienced by this high-risk population, a novel adaptation of the evidence-based DSME model and subsequent testing in a community-based setting are needed.

Using a Community Based Participatory Research (CBPR) approach, we have conducted four focus groups and individual interviews with the Marshallese community to better understand how to best address the well-established need for diabetes education. Through interviews and focus groups, Marshallese participants pointed out that the delivery method and the concept of self-management as an individual experience are problematic components. DSME was designed with a very Western societal approach, which is highly individualistic. The Marshallese have a highly collectivist culture and the idea of -self‖ management is counter to their cultural values. As stakeholders described, -we eat together from one pot. For one person to refuse the food from that one pot is not just inconvenient, it is shameful. It shames the person and the person's family. It is not an acceptable option. We will not do it. The interviewees stated that any changes must be a family change. Incorporating collectivist and family concepts into the delivery mechanism is imperative. Through the interviews and focus groups, the Marshallese community suggested that DSME be implemented within a family model with a family group receiving DSME so that the entire family can benefit and the patient can be supported in their effort to make lifestyle changes. Because ~30-50% of the Marshallese community have type 2 diabetes, this approach could be even more beneficial.

Hypothesis and/or Specific Aims or Objectives

We hypothesize that a culturally adapted DSME implemented in a family model will result in better diabetes management outcomes compared with standard DSME for the Marshallese.

In the family delivery model, a participant is encouraged to invite his/her family members to the diabetes educational sessions. As outlined by stakeholders, the model has several potential benefits. First, patients are empowered to invite the people they define as family and as appropriate for taking part in the sessions with them. Second, the education will engage the patient-defined support unit. Third, given the high-rate of diabetes within the community, it is highly probable that others within the group will have Type 2 diabetes or pre-diabetes and may benefit from the intervention as well.

Our aim is to test an Adapted DSME using a mixed-methods approach. Marshallese participants with type 2 diabetes will be recruited. Those who are assigned to the family model will be asked to invite one to ten adult members of their families to participate in the DSME. Given that ~30-50% of adults in the Marshallese community have type 2 diabetes, and the Marshallese typically have large families, recruitment for this nontraditional model is plausible. Furthermore, the method was designed from input from our CBPR partnership with the Marshallese.

This research is highly translational. It will help bridge the gap between knowledge of an effective DSME intervention and actual implementation of the intervention among a Pacific Islander population with especially high rates of type 2 diabetes and significant health disparities.

ELIGIBILITY:
Inclusion Criteria:

Primary Participant:

* Must be 18 years or older
* Self-reported Diabetes Mellitus Type 2 diagnosis by a health care provider
* Self-reported Marshallese ethnicity or descent

Secondary (Family) Participant:

* Must be 18 years or older

Exclusion Criteria:

* Younger than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2015-06; Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter O Kohler, M.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences Northwest, Fayetteville, Arkansas, United States

REFERENCES:
- [Derived] Felix HC, Narcisse MR, Long CR, McElfish PA. Effects of a family diabetes self-management education intervention on the patients' supporters. Fam Syst Health. 2020 Jun;38(2):121-129. doi: 10.1037/fsh0000470. Epub 2020 Apr 13. PMID 32281816
- [Derived] McElfish PA, Purvis RS, Scott AJ, Haggard-Duff LK, Riklon S, Long CR. "The results are encouragements to make positive changes to be healthier:" qualitative evaluation of Marshallese participants' perceptions when receiving study results in a randomized control trial. Contemp Clin Trials Commun. 2020 Feb 19;17:100543. doi: 10.1016/j.conctc.2020.100543. eCollection 2020 Mar. PMID 32140610
- [Derived] McElfish PA, Long CR, Kohler PO, Yeary KHK, Bursac Z, Narcisse MR, Felix HC, Rowland B, Hudson JS, Goulden PA. Comparative Effectiveness and Maintenance of Diabetes Self-Management Education Interventions for Marshallese Patients With Type 2 Diabetes: A Randomized Controlled Trial. Diabetes Care. 2019 May;42(5):849-858. doi: 10.2337/dc18-1985. Epub 2019 Mar 12. PMID 30862659

RESULTS

PARTICIPANT FLOW:
Period: Immediate Post-intervention
Arm/Group | Adapted DSME | Standard DSME
Started | 110 | 111
Completed | 107 | 101
Not Completed | 3 | 10
Period: 6 Months Post-intervention
Arm/Group | Adapted DSME | Standard DSME
Started (All participants were recontacted whether or not they completed post-intervention data collection.) | 107 | 101
Completed | 96 | 92
Not Completed | 11 | 9
Period: 12 Months Post-intervention
Arm/Group | Adapted DSME | Standard DSME
Started (All participants were recontacted whether or not they completed previous data collection events.) | 96 | 92
Completed | 83 | 90
Not Completed | 13 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adapted DSME | Standard DSME | Total
Number analyzed (Participants) | 110 | 111 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (11.1) | 53.0 (10.6) | 52.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 72 | 130
  Male | 52 | 39 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 110 | 111 | 221
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 110 | 111 | 221
HbA1c (%) (unadjusted) [Mean (Standard Deviation); unit: Percent Glycated Hemoglobin (unadjusted)] | 10.51 (2.37) | 10.41 (2.22) | 10.46 (2.29)

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control, Measured by Change in Adjusted Mean HbA1c (%) From Baseline to Immediate Post-intervention, 6 Months Post-intervention, and 12 Months Post-intervention.
Description: A Siemens analyzer (point of care) was utilized to calculate HbA1c levels for each participant. The primary outcome measure was change in adjusted mean HbA1c (%) from baseline to immediate post-intervention, 6 months post-intervention, and 12 months post-intervention. Analyses were adjusted for baseline sex, age, education, marital status, employment status, use of diabetes medication, and households containing multiple participants. The mean HbA1c values presented here have been adjusted, whereas the mean HbA1c values presented in the Baseline Data section are unadjusted.
Time Frame: Baseline, Immediate post-intervention, 6 months post-intervention, 12 months post-intervention
Measure: Mean (95% Confidence Interval); unit: Percent Glycated Hemoglobin (adjusted)
Arm/Group | Adapted DSME | Standard DSME
Number analyzed (Participants) | 110 | 111
Percent Glycated Hemoglobin (adjusted)
  Baseline | 10.48 [10.08 to 10.89] | 10.46 [10.07 to 10.86]
  Immediate post-intervention | 9.30 [8.90 to 9.70] | 9.91 [9.50 to 10.32]
  6 months post-intervention | 9.81 [9.40 to 10.23] | 10.26 [9.84 to 10.68]
  12 months post-intervention | 9.61 [9.17 to 10.04] | 10.38 [9.96 to 10.81]
Statistical Analysis 1: Comparison: Adapted DSME vs Standard DSME; The outcome variable for these analyses is Change in mean HbA1c from baseline to immediate post-intervention, 6 months post-intervention, and 12 months post-intervention; Test type: Superiority; p = 0.038, Linear mixed effects regression — The p-value above reflects results of between-arms analysis of mean change in HbA1c from baseline to immediate post-intervention. 6 months between-arms p-value = 0.139; 12 months between-arms p-value = 0.013. Analyses do not include imputed values; Adjusted for baseline sex, age, education, marital status, employment, use of diabetes medication, and households containing multiple participants

2. Secondary Outcome: Change in Mean BMI From Baseline to Immediate Post-intervention, 6 Months Post-intervention, and 12 Months Post-intervention
Description: Participant weight (without shoes) was measured in light clothing to the nearest 0.5 lb (0.2 kg) using a calibrated digital scale. Height (without shoes) was measured to the nearest 0.5 cm using a stadiometer. Weight and height were used to compute a continuous measure of BMI (kg/m²).
Time Frame: Baseline, Immediate post-intervention; 6 months post-intervention; 12 months post-intervention
Measure: Mean (95% Confidence Interval); unit: BMI (kg/m²)
Arm/Group | Adapted DSME | Standard DSME
Number analyzed (Participants) | 110 | 111
BMI (kg/m²)
  Baseline | 30.58 [29.60 to 31.55] | 31.46 [30.50 to 32.42]
  Immediate post-intervention | 30.66 [29.68 to 31.63] | 31.49 [30.53 to 32.46]
  6 months post-intervention | 30.97 [29.99 to 31.95] | 31.39 [30.42 to 32.36]
  12 months post-intervention | 30.78 [29.80 to 31.77] | 31.32 [30.35 to 32.29]
Statistical Analysis 1: Comparison: Adapted DSME vs Standard DSME; The outcome variable for these analyses is Change in mean BMI from baseline to immediate post-intervention, 6 months post-intervention, and 12 months post-intervention; Test type: Superiority; p = 0.234, Linear mixed effects regression — The p-value above reflects results of between-arms analysis of change in mean BMI from baseline to immediate post-intervention. 6 months between-arms p-value = 0.552; 12 months between-arms p-value = 0.447. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Change in Mean Total Cholesterol (mg/dL) From Baseline to Immediate Post-intervention, 6 Months Post-intervention, and 12 Months Post-intervention.
Description: Through finger prick blood collection, point of care tests were used to test fasting lipids using a commercial lipid panel kit and Cholestech LDX analyzer. Analyses were adjusted for baseline sex, age, education, marital status, employment status, use of diabetes medication, and households containing multiple participants.
Time Frame: Baseline, Immediate post-intervention, 6 months post-intervention, 12 months post-intervention
Measure: Mean (95% Confidence Interval); unit: Total Cholesterol (mg/dL)
Arm/Group | Adapted DSME | Standard DSME
Number analyzed (Participants) | 110 | 111
Total Cholesterol (mg/dL)
  Baseline | 181.39 [174.25 to 188.52] | 189.08 [181.97 to 196.19]
  Immediate post-intervention | 170.15 [162.92 to 177.37] | 182.64 [175.35 to 189.94]
  6 months post-intervention | 178.69 [171.27 to 186.12] | 175.84 [168.30 to 183.37]
  12 months post-intervention | 170.88 [163.15 to 178.61] | 180.79 [173.24 to 188.34]
Statistical Analysis 1: Comparison: Adapted DSME vs Standard DSME; The outcome variable for these analyses is Change in mean Total Cholesterol (mg/dL) from baseline to immediate post-intervention, 6 months post-intervention, and 12 months post-intervention; Test type: Superiority; p = 0.019, Linear mixed effects regression — The p-value above reflects results of between-arms analysis of change in mean total chol from baseline to immediate post-intervention. 6 months between-arms p-value=0.598; 12 months between-arms p-value=0.073. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Change in Mean High-density Lipoproteins (HDL) From Baseline to Immediate Post-intervention, 6 Months Post-intervention, and 12 Months Post-intervention.
Description: A commercial lipid panel kit and Cholestech LDX analyzer were used to assess HDL levels. The outcome measure was change in mean HDL from baseline to immediate post-intervention, 6 months post-intervention, and 12 months post-intervention. Analyses were adjusted for baseline sex, age, education, marital status, employment status, use of diabetes medication, and households containing multiple participants.
Time Frame: Baseline, Immediate post-intervention, 6 months post-intervention, 12 months post-intervention
Measure: Mean (95% Confidence Interval); unit: HDL (mg/dL)
Arm/Group | Adapted DSME | Standard DSME
Number analyzed (Participants) | 110 | 111
HDL (mg/dL)
  Baseline | 36.43 [34.47 to 38.39] | 36.99 [35.04 to 38.93]
  Immediate post-intervention | 37.53 [35.56 to 39.50] | 35.63 [33.63 to 37.63]
  6 months post-intervention | 39.34 [37.31 to 41.36] | 35.49 [33.46 to 37.52]
  12 months post-intervention | 37.50 [35.39 to 39.60] | 35.58 [33.53 to 37.62]
Statistical Analysis 1: Comparison: Adapted DSME vs Standard DSME; The outcome variable for these analyses is Change in mean HDL (mg/dL) from baseline to immediate post-intervention, 6 months post-intervention, and 12 months post-intervention; Test type: Superiority; p = 0.186, Linear mixed effects regression — The p-value above reflects results of between-arms analysis of mean change in HDL from baseline to immediate post-intervention. 6 months between-arms p-value=0.009; 12 months between-arms p-value=0.201. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Change in Probability of Performing Diabetes Self-care Behaviors From Baseline to 12 Months Post-intervention: Check Blood Glucose Daily
Description: This measure assesses whether or not each participant reported checking her/his blood glucose at least daily at baseline and 12 months post-intervention. This measure of participant-reported current level of diabetes self-care was assessed through an item from the Behavioral Risk Factor Surveillance System (BRFSS) Diabetes Module. (Because three of the diabetes self-care behaviors we assessed are expected to occur annually (e.g., annual doctor visit), analyses of self-care behaviors focus on change from baseline to 12 months post-intervention to allow for a year to elapse between time points.)
Time Frame: Baseline, 12 months post-intervention
Measure: Mean (95% Confidence Interval); unit: Probability
Arm/Group | Adapted DSME | Standard DSME
Number analyzed (Participants) | 110 | 111
Probability
  Baseline probability | 0.44 [0.31 to 0.57] | 0.53 [0.39 to 0.65]
  12 months probability | 0.94 [0.85 to 0.98] | 0.82 [0.70 to 0.90]
Statistical Analysis 1: Comparison: Adapted DSME vs Standard DSME; To facilitate interpretation of regression coefficients, estimates obtained in the logit scale (log odds) were transformed into probability scale; Test type: Superiority; p = 0.040, Mixed effects logistic regression — The p-value above represents results of analysis of the between-arm changes in probability of performing the self-care behavior from baseline to 12 months post-intervention. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Change in Probability of Performing Diabetes Self-care Behaviors From Baseline to 12 Months Post-intervention: Seen Doctor or Other Health Professional in Past 12 Months for Diabetes
Description: This measure assesses whether or not each participant reported seeing a doctor, nurse, or other health professional for her/his diabetes within the past 12 months at baseline and 12 months post-intervention. This measure of participant-reported current level of diabetes self-care was assessed through an item from the Behavioral Risk Factor Surveillance System (BRFSS) Diabetes Module. (Because three of the diabetes self-care behaviors we assessed are expected to occur annually (e.g., annual doctor visit), analyses of self-care behaviors focus on change from baseline to 12 months post-intervention to allow for a year to elapse between time points.)
Time Frame: Baseline, 12 months post-intervention
Measure: Mean (95% Confidence Interval); unit: Probability
Arm/Group | Adapted DSME | Standard DSME
Number analyzed (Participants) | 110 | 111
Probability
  Baseline probability | 0.77 [0.66 to 0.85] | 0.82 [0.72 to 0.89]
  12 months probability | 0.92 [0.84 to 0.96] | 0.88 [0.79 to 0.93]
Statistical Analysis 1: Comparison: Adapted DSME vs Standard DSME; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.312, Mixed Effects Logistic Regression — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: Change in Probability of Performing Diabetes Self-care Behaviors From Baseline to 12 Months Post-intervention: Foot Exam by Doctor or Other Health Professional in Past 12 Months
Description: This measure assesses whether or not each participant reported having a health professional check her/his feet for any sores or irritations in the past 12 months at baseline and 12 months post-intervention. This measure of participant-reported current level of diabetes self-care was assessed through an item from the Behavioral Risk Factor Surveillance System (BRFSS) Diabetes Module. (Because three of the diabetes self-care behaviors we assessed are expected to occur annually (e.g., annual doctor visit), analyses of self-care behaviors focus on change from baseline to 12 months post-intervention to allow for a year to elapse between time points.)
Time Frame: Baseline, 12 Months Post-Intervention
Measure: Mean (95% Confidence Interval); unit: Probability
Arm/Group | Adapted DSME | Standard DSME
Number analyzed (Participants) | 110 | 111
Probability
  Baseline probability | 0.49 [0.39 to 0.59] | 0.47 [0.37 to 0.57]
  12 months probability | 0.53 [0.42 to 0.64] | 0.49 [0.38 to 0.60]
Statistical Analysis 1: Comparison: Adapted DSME vs Standard DSME; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.622, Mixed effects logistic regression — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 1, analysis 1]

8. Secondary Outcome: Change in Probability of Performing Diabetes Self-care Behaviors From Baseline to 12 Months Post-intervention: Eye Exam in Past 12 Months
Description: This measure assesses whether or not each participant reported having an eye exam in which the pupils were dilated in the past 12 months at baseline and 12 months post-intervention. This measure of participant-reported current level of diabetes self-care was assessed through an item from the Behavioral Risk Factor Surveillance System (BRFSS) Diabetes Module. (Because three of the diabetes self-care behaviors we assessed are expected to occur annually (e.g., annual doctor visit), analyses of self-care behaviors focus on change from baseline to 12 months post-intervention to allow for a year to elapse between time points.)
Time Frame: Baseline, 12 Months Post-Intervention
Measure: Mean (95% Confidence Interval); unit: Probability
Arm/Group | Adapted DSME | Standard DSME
Number analyzed (Participants) | 110 | 111
Probability
  Baseline probability | 0.35 [0.26 to 0.46] | 0.34 [0.25 to 0.44]
  12 months probability | 0.41 [0.30 to 0.53] | 0.41 [0.30 to 0.52]
Statistical Analysis 1: Comparison: Adapted DSME vs Standard DSME; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.957, Mixed effects logistic regression — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 1, analysis 1]

9. Secondary Outcome: Change in Probability of Performing Diabetes Self-care Behaviors From Baseline to 12 Months Post-intervention: Maintain a Normal Weight
Description: This measure assesses whether or not each participant had a normal weight at baseline and 12 months post-intervention as indicated by body mass index (i.e., body mass index between 18.5 to 24.9). Participant weight (without shoes) was measured in light clothing to the nearest 0.5 lb (0.2 kg) using a calibrated digital scale. Height (without shoes) was measured to the nearest 0.5 cm using a stadiometer. Weight and height were used to compute a continuous measure of BMI (kg/m²). (Because three of the diabetes self-care behaviors we assessed are expected to occur annually (e.g., annual doctor visit), analyses of self-care behaviors focus on change from baseline to 12 months post-intervention to allow for a year to elapse between time points.)
Time Frame: Baseline, 12 Months Post-Intervention
Measure: Mean (95% Confidence Interval); unit: Probability
Arm/Group | Adapted DSME | Standard DSME
Number analyzed (Participants) | 110 | 111
Probability
  Baseline probability | 0.14 [0.09 to 0.23] | 0.07 [0.03 to 0.13]
  12 months probability | 0.14 [0.08 to 0.24] | 0.08 [0.04 to 0.15]
Statistical Analysis 1: Comparison: Adapted DSME vs Standard DSME; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.147, Mixed effects logistic regression — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 1, analysis 1]

10. Secondary Outcome: Change in Probability of Performing Diabetes Self-care Behaviors From Baseline to 12 Months Post-intervention: Engage in Recommended Level of Physical Activity
Description: This measure assesses whether or not each participant reported engaging in 60 minutes or more of vigorous activity per week or 150 minutes or more of moderate activity per week at baseline and 12 months post-intervention. This measure was lightly adapted from the measure of physical activity used here: L. Jiang, S. Chen, B. Zhang, J. Beals, C.M. Mitchell, S.M. Manson, et al. Longitudinal patterns of stages of change for exercise and lifestyle intervention outcomes: an application of latent class analysis with distal outcomes. Prev. Sci., 17 (2016), pp. 398-409. (Because three of the diabetes self-care behaviors we assessed are expected to occur annually (e.g., annual doctor visit), analyses of self-care behaviors focus on change from baseline to 12 months post-intervention to allow for a year to elapse between time points.)
Time Frame: Baseline, 12 Months Post-Intervention
Measure: Mean (95% Confidence Interval); unit: Probability
Arm/Group | Adapted DSME | Standard DSME
Number analyzed (Participants) | 110 | 111
Probability
  Baseline probability | 0.09 [0.05 to 0.16] | 0.04 [0.02 to 0.10]
  12 months probability | 0.09 [0.04 to 0.17] | 0.05 [0.02 to 0.12]
Statistical Analysis 1: Comparison: Adapted DSME vs Standard DSME; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.326, Mixed effects logistic regression — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 1, analysis 1]

11. Secondary Outcome: Change in Mean Fasting Glucose From Baseline to Immediate Post-intervention, 6 Months Post-intervention, and 12 Months Post-intervention
Description: Informally and in response to a survey item, many participants reported that they had not adhered to instructions to fast before data collection. For this reason, we were unable to collect valid measures for fasting glucose, low-density lipoproteins (LDL), and triglycerides.
Time Frame: Baseline, Immediate Post-Intervention, 6 Months Post-Intervention, 12 Months Post-Intervention
Reporting Status: Not Posted

12. Secondary Outcome: Change in Mean Low-density Lipoproteins (LDL) From Baseline to Immediate Post-intervention, 6 Months Post-intervention, and 12 Months Post-intervention
Description: as for outcome 11
Time Frame: Baseline, Immediate Post-Intervention, 6 Months Post-Intervention, 12 Months Post-Intervention
Reporting Status: Not Posted

13. Secondary Outcome: Change in Mean Triglycerides From Baseline to Immediate Post-intervention, 6 Months Post-intervention, and 12 Months Post-intervention
Description: as for outcome 11
Time Frame: Baseline, Immediate Post-Intervention, 6 Months Post-Intervention, 12 Months Post-Intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From enrollment to 1 year, 4 months post-enrollment
Description: Study staff assessed presence of adverse events via regular contact with participants from both study arms throughout the duration of the study.
Groups:
- Family Model DSME: Participants assigned to this arm received an intervention that includes culturally-adapted DSME with their participating family members in a family/home setting.
Arm/Group | Standard DSME | Family Model DSME
All-Cause Mortality (participants affected / at risk) | 1/111 | 3/110
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/110
Other Adverse Events (participants affected / at risk) | 0/111 | 0/110

LIMITATIONS AND CAVEATS:
We were unable to collect valid measures for fasting glucose, low-density lipoproteins (LDL), and triglycerides, as participants reported they had not adhered to instructions to fast before data collection events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT02407132/Prot_SAP_000.pdf